CLINICAL TRIAL: NCT06874790
Title: Randomized Controlled Trial of a Choice-driven, Interactive, Storytelling Web-based App to Investigate Mental Health Treatment Initiation Among Symptomatic Latinas
Brief Title: RCT for Latina Mental Health Using Web-Based Apps
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, MarySue Heilemann, PhD, RN, FAAN, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 24-5962; R01MH137232 (NIH)
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Mental Health; Anxiety; Depression; Well-Being, Psychological
Keywords: Latina; Women; Therapy
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Individual-level randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catalina transmedia web-based app (Experimental): Access to Confronting My Emotions/ Enfrentando Mis Emociones (Catalina), an interactive web-based app containing 31 minutes of story based, character-driven videos, featuring evidence-informed Latina characters (Catalina and Veronica) in a relatable story about dealing with depression and anxiety. All features are available 24 hours/day in Spanish and English via a participant's unique link, including access to "Veronica's Blog" linked to the story, and links to resources such as infographics on depression and anxiety, hotlines and helplines, free evidence-based apps, online support groups, SAMHSA's MH service locator plus "Veronica's" recommendation of up to 3 Latinx-serving MH Tx clinics in LA & Orange Counties where participants can see a primary care physician for referral to MH therapy or pharmacotherapy. Monthly text/email messages will be sent for 9 months to prompt/remind Latinas they can use their unique link to re-watch videos and re-visit Veronica's blog.
  Interventions: Behavioral: Catalina
- Links to informational videos (Active Comparator): Access to the control web-based app that offers links to 31 minutes of publicly available informational videos specifically about depression and anxiety in Spanish and English (that are not story based and feature no fictionalized characters), available 24 hours/ day via participant's unique link on Chorus. It will provides direct links to 3 public websites: 1) Mental Health America, 2) Anxiety & Depression Association of America, 3) SAMHSA. All offer even more links to various MH resources, platforms, videos, and to SAMHSA's MH service locator by ZIP Code including to low cost sites for MH Tx.
  Interventions: Behavioral: Control webpage

INTERVENTIONS:
Behavioral: Catalina — Catalina transmedia web-based app intervention with 10 story-based videos (including bonus story extender videos) totaling 31 minutes plus the blog of the character, "Veronica," which has MH resource links including Veronica's recommendations of at least 3 local Latinx-serving clinics in LA and Orange County ZIP Codes that offer low-cost MH Tx.
  Other Names: Confronting My Emotions; Enfrentando Mis Emociones
  Arms: Catalina transmedia web-based app
Behavioral: Control webpage — Links to informational videos (totaling 31 minutes) on depression and anxiety, listing of the same 3 local Latinx-serving clinics in LA and Orange County ZIP codes that offer low-cost MH Tx, and links to nationally available websites that offer resources (including access to service locators).
  Arms: Links to informational videos

SUMMARY:
This study compares a choice-driven, interactive, evidence-informed storytelling web-based app intervention with links to resources and treatment (Tx) recommendations (made by a character via her blog) and Tx locator, to a web-based app with links to publicly available informational internet videos, MH resources, and a treatment locator for at least moderately anxious/depressed untreated English and Spanish speaking Latinas to determine if a story-based, character-driven approach is more effective for catalyzing mental health treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Latina (women who are from or have family ties to Latin America)
* Currently resides in LA or Orange County
* Age 18 and older
* Able to speak, read, and write in English or Spanish
* Score 10 or higher on GAD-7 and/or PHQ-8
* Access to the internet via smartphone, tablet, or computer
* Not currently receiving mental health therapy or pharmacotherapy
* Has not accessed mental health services during the previous 6 months

Exclusion Criteria:

* Not Latina or Hispanic
* Under age 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Screening is based on self-identification as woman or female
Enrollment: 700 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Initiating Mental Health Treatment (MH Tx) | 9 months
  MH Tx initiation, defined as completing a MH specialist visit (initial evaluation or therapy visit) or a primary care visit that results in a pharmacotherapy prescription as documented by EHR data at the site identified by the participant as where they initiated MH Tx.

SECONDARY OUTCOMES:
Psychological openness | 9 months
  Psychological openness (attitudes) subscale score of the Inventory of Attitudes towards Seeking Mental Health Services (IASMHS). The IASMHS is a 24 item scale and has three internally consistent factors: psychological openness, help-seeking propensity, and indifference to stigma. The subscales,range from 0 to 32. Higher scores indicate more positive attitude toward seeking mental health services.
Mental health help seeking attitude | 9 months
  The Mental Health Seeking Attitudes Scale (MHSAS) contains 9 items which produce a single mean score, ranging 1-7. It measures respondents' overall evaluation (unfavorable vs. favorable) of their seeking help from a mental health professional if they found themselves to be dealing with a mental health concern. A higher score indicates a more favorable attitude toward seeking help.
Propensity to seek help | 9 months
  Help seeking propensity subscale score of the Inventory of Attitudes towards Seeking Mental Health Services (IASMHS). The IASMHS is a 24 item scale and has three internally consistent factors: psychological openness, help-seeking propensity, and indifference to stigma. Subscales range from 0 to 32. Higher scores indicate a greater willingness to seek help.
Indifference to Stigma | 9 months
  Indifference to Stigma subscale score of the Inventory of Attitudes towards Seeking Mental Health Services (IASMHS). The IASMHS is a 24 item scale and has three internally consistent factors: psychological openness, help-seeking propensity, and indifference to stigma. The subscale contains 8 items related to how concerned an individual would feel if others knew they were seeking psychological help, with each item rated on a 5-point Likert scale from 0 (disagree) to 4 (agree); a higher score indicates a greater indifference to stigma; meaning the person is less concerned about others finding out about their mental health treatment.
Stigma Concerns | 9 months
  Stigma Concerns about Care (SCC) is a 3-item questionnaire with responses on a 1-10 point scale, with higher scores indicating more concern about stigma.

OTHER OUTCOMES:
Depression | 9 months
  The Patient Health Questionnaire 8 (PHQ-8) is an 8 item questionnaire for depression symptoms experienced during the preceding 2 weeks. Responses are scaled 0-3, total score range 0-24. A score of 10 or greater is considered major depression, 20 or more is severe major depression.
Anxiety | 9 months
  The Generalized Anxiety Disorder-7 (GAD7) is a 7-item questionnaire to measure the severity of anxiety over the preceding 2 weeks. Responses range from 0 (not at all) to 3 (nearly every day), with total score range 0-21. Higher scores indicate more severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: MarySue V. Heilemann, PhD,RN,FAAN, Principal Investigator — UCLA School of Nursing
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No